CLINICAL TRIAL: NCT04508907
Title: Pilot Study for the Use of Shortened Preemptive Therapy With Glecaprevir/Pibrentasvir (G/P) and Ezetimibe in Hepatitis C Seronegative Solid Organ Transplant Recipients (Kidney, Heart, Lung and/or Pancreas) of Hepatitis C Viremic Donors
Brief Title: A Study to Evaluate Preemptive Therapy in Hepatitis C (HCV) Organ Transplant Recipients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bashar Aqel, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-001964
Record Dates: First submitted 2020-07-30; First posted 2020-08-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis C; Kidney Transplant; Complications; Heart Transplant Infection
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir and pibrentasvir; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1: Pre-emptive Treatment Arm (Experimental): Single arm study were all recipients of HCV viremic organs will receive combination therapy.
  Interventions: Drug: Mavyret

INTERVENTIONS:
Drug: Mavyret — Mavyret and Zetia for 8 days to prevent HCV infection in solid organ recipients
  Other Names: Zetia

SUMMARY:
This study is being done to determine the effectiveness of using a combination of two different drugs in preventing the transmission of HCV from a HCV positive donor to a HCV negative solid organ recipient.

ELIGIBILITY:
Inclusion criteria:

* Listed kidney, heart, lung and/or pancreas patients who are negative for chronic hepatitis C infection
* Willing to accept and consent for accepting hepatitis C positive graft

Exclusion criteria:

* Existing chronic liver disease (liver cirrhosis)
* Concomitant infection with HIV or Chronic hepatitis B
* Patient or any member of patient family or care giver team who does not understand or accept the risk of an acquired HCV infection
* Pregnancy (Pregnant patients do not undergo solid organ transplants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of prevention of HCV viremia in recipients of HCV viremic solid organs | 3 months
  The study will assess the percentage of patient who will not become HCV viremic using this preemptive treatment protocol.
Graft and patient survival | 1 year
  Study will assess the overall 1 year patient and graft survival.

CONTACTS AND LOCATIONS:
Overall Officials: Bashar A Aqel, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials